CLINICAL TRIAL: NCT01387633
Title: Educational Intervention and Social Support in Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: University of São Paulo, University of Sao Paulo at Ribeirão Preto College of Nursing
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: diabetes2011
Record Dates: First submitted 2011-06-16; First posted 2011-07-04 (Estimated); Last update posted 2011-07-04 (Estimated); Status verified 2010-02

CONDITIONS: Diabetes Mellitus
Keywords: Nursing care; Diabetes mellitus; Health Education; Patient compliance; Social support; Self-efficacy; Adaptation strategy
MeSH Terms: conditions — Diabetes Mellitus; Health Education; Patient Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Educational intervention through telephone contact (Experimental): Educational intervention for family members/caregivers of people with diabetes mellitus through telephone contact
  Interventions: Other: Educational intervention for family members/caregivers of people with diabetes mellitus through telephone contact
- Educational intervention group (Active Comparator): Educational intervention group for people with diabetes through Diabetes Conversation Maps.
  Interventions: Other: Educational intervention group for people with diabetes through Diabetes Conversation Maps

INTERVENTIONS:
Other: Educational intervention for family members/caregivers of people with diabetes mellitus through telephone contact — For family members/caregivers: telephone contacts will be conducted in day and time which family member/caregiver prefers, and he/she may make collect calls to the researcher always he/she judges it necessary during the period of study. Phone contacts will be recorded to ensure the registration of orientation given, using a digital phone recorder PCTEL. And they will be arranged with the technique of motivational interviewing that includes the skills to ask, listen and inform. For this, protocols based on these skills, which the covered topics will be those worked in group sessions through Diabetes Conversation Maps. Voice quality related to the tone, volume and clarity as well as the skills and strategies to listen to the interviews will be worked under the guidance of an audiologist
  Arms: Educational intervention through telephone contact
Other: Educational intervention group for people with diabetes through Diabetes Conversation Maps — For people with diabetes mellitus: educational interventions will be conducted in accordance with the assumptions of the Social Cognitive Theory, through Diabetes Conversation Maps , whose use is consistent with this theory (ADA, 2007). Diabetes Conversation Maps are a tool which involves people in the learning process about the disease, to make them able to process information more effectively and use them in making daily decisions in the management of diabetes mellitus (DM). It is recommended that this tool is used in small groups of three to ten people, in order to provide dynamic discussions among the participants (ADA, 2007). Currently, the maps that cover the following learning contexts: How the Body and Diabetes Work, Healthy Eating and Physical Activity, and Medication Treatment and Monitoring of Blood Glucose; Achieving the Goals with the Insulin and Weather Map of Diabetic Foot are available for the Brazilian Portuguese language.
  Arms: Educational intervention group

SUMMARY:
The purpose of this study is to evaluate the impact of an educational program for people with diabetes mellitus based on the family social support.

DETAILED DESCRIPTION:
H0: The person with diabetes who participates in the educational group whose family member/caregiver receives educational interventions hasn't greater glycemic control.

HA: The person with diabetes who participates in the educational group whose family member/caregiver receives educational interventions has greater glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* People with DM2
* Both sexes
* Minimum age of 40 years
* Able to dialogue
* Lack of complications in advanced

Exclusion Criteria:

* Hemodialysis treatment
* Amaurosis
* Sequelae of Stroke and/or Heart Failure
* Previous amputations at any level of the lower limb
* Active ulcer in the lower limbs
* People in wheelchairs and/or litter
* People with limited understanding of the instruments due to cultural factors

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2011-06; Primary Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
glycated hemoglobin | 21 mounths
fasting plasma glucose | 21 mounths
triglycerides | 21 mounths
total cholesterol and fractions | 21 mounths
microalbuminuria | 21 mounths
urea | 21 mounths
creatinine | 21 mounths
body mass index | 21 mounths
waist circumference | 21 mounths
blood pressure | 21 mounths

SECONDARY OUTCOMES:
Perceived Self-Efficacy: Diabetes Management Self-efficacy Scale for Patients with Type 2 Diabetes Mellitus | 21 mounths
Knowledge about diabetes mellitus: Diabetes Mellitus knowledge (DKN-A) | 21 mounths
Adherence to medication treatment: Self-Reported Measure of Medication Adherence (Measure of Treatment Adherence - MTA) | 21 mounths
Adherence to self care: Summary of Diabetes Self-Care Activities Questionnaire (SDSCA) ( Diabetes Self-Care Activities Questionnaire) | 21 mounths
Perception of stress: Perceived Stress Scale (Perceived Stress Scale) | 21 mounths
Ways of coping: Ways of Coping Scale (Ways of Coping Scale) | 21 mounths
Acceptance of Illness (Acceptance of Illness Scale) | 21 mounths
Perception of social support: The Social Support Network Inventory | 21 mounths
Self-monitoring of blood glucose | 21 mounths

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo, Ribeirão Preto, São Paulo, Brazil